CLINICAL TRIAL: NCT05341219
Title: Effect of Light Needle in the Treatment of Opioid Use Disorder: A Randomized Controlled Trial
Brief Title: Light Needle for Opioid Use Disorder
Acronym: OUD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Kaohsiung Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMRPG8M0031; MOHW111-CMAP-M-113-112103 (Other Grant/Funding Number: The Ministry of Health and Welfare); MOHW112-CMAP-M-113-000005-C (Other Grant/Funding Number: The Ministry of Health and Welfare)
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Opioid Use Disorder
Keywords: Light needle; Opioid use disorder; Heroin addiction; Methadone maintenance treatment; Traditional Chinese medicine
MeSH Terms: conditions — Opioid-Related Disorders; Heroin Dependence

STUDY DESIGN:
Intervention Model Description: Subjects recruited from the two institutions are being randomly allocated to the experimental group (light needle plus methadone maintenance treatment, n = 50, expected), or the control group (light needle without laser output plus methadone maintenance treatment, n = 50, expected). The study participants will receive 12 sessions of light needle therapy within 4 weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation concealment was implemented through the use of numbered containers. The allocation sequence was concealed from the researcher enrolling and assessing participants in sequentially numbered, opaque, sealed, and stapled envelopes. The trial participants, outcome assessors, and data analysts will be blinded after assignment to interventions using label A and B for the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- light needle therapy (Experimental): The study participants will receive 12 sessions of light needle therapy within 4 weeks using a gallium aluminum arsenide Physiolaser olympic (maximal power, 60mW; wavelength, 655 nm; area of probe, 0.008 cm2; power density, 7.5 W/cm2; pulsed-wave; RJ-Laser, Reimers & Janssen GmbH, Waldkirch, Germany). Those in the experimental group received a total 135 J of energy delivered from 6 light needles being placed between LU7 and LU9. The light needle therapy was applied to each point for 15 min.
  Interventions: Procedure: Light needle therapy
- sham light needle therapy (Sham Comparator): The study participants will receive 12 sessions of sham light needle therapy, without any laser output (no stimulation), within 4 weeks using a gallium aluminum arsenide Physiolaser olympic. Those in the control group received 0 J of energy delivered from 6 light needles being placed between LU7 and LU9 for 15 min.
  Interventions: Procedure: Sham light needle therapy

INTERVENTIONS:
Procedure: Light needle therapy — The study participants will receive 12 sessions of light needle therapy within 4 weeks using a gallium aluminum arsenide Physiolaser olympic (maximal power, 60mW; wavelength, 655 nm; area of probe, 0.008 cm2; power density, 7.5 W/cm2; pulsed-wave; RJ-Laser, Reimers & Janssen GmbH, Waldkirch, Germany). Those in the experimental group received a total 135 J of energy delivered from 6 light needles being placed between LU7 and LU9. The light needle therapy was applied to each point for 15 min.
  Arms: light needle therapy
Procedure: Sham light needle therapy — The study participants will receive 12 sessions of sham light needle therapy, without any laser output (no stimulation), within 4 weeks using a gallium aluminum arsenide Physiolaser olympic. Those in the control group received 0 J of energy delivered from 6 light needles being placed between LU7 and LU9 for 15 min.
  Arms: sham light needle therapy

SUMMARY:
This randomized-controlled study investigates the effect of adjuvant light needle in the treatment of heroin addicts. One hundred heroin addicts older than 20 years old enrolled from the Addiction Treatment Center at Kaohsiung Chang Gung Memorial Hospital and Department of Psychiatry at Kaohsiung Medical University Hospital are randomly allocated to experimental or control group. Subjects in experimental group are treated with light needle on the wrist pulse (Cunkou) 12 times within 4 weeks. Subjects in the control group received a sham light needle treatment, without any laser output. Outcome measurements include check of urine morphine, report of the subjects' times or days of heroin use, self-filling Visual Analogue Scales of heroin craving / refusal of heroin use (0-10 points) during last week, report of the subjects' quality of life using Short Form-12v2, and record of the subject's pulse diagnosis and heart rate variability before and after treatment.

DETAILED DESCRIPTION:
Background: Heroin addiction remains a significant public health problem worldwide, and relapse to heroin use following cessation of agonist maintenance treatment is common. The problems associated with use of opioid agonists mean that non-opioid therapies need to be developed to ameliorate acute and protracted opioid withdrawal syndromes.

Objective: To investigate the effect of adjuvant light needle therapy in patients with opioid use disorder on methadone maintenance treatment.

Methods: One hundred participants with opioid use disorder on methadone maintenance treatment will be enrolled from the addiction treatment center at Kaohsiung Chang Gung Memorial Hospital and Department of Psychiatry at Kaohsiung Medical University Hospital, and randomly allocated to the experimental or control group. The experimental group is receiving 12 sessions of light needle therapy within 4 weeks. The control group is receiving sham light needle treatment, without any laser output. Urinary morphine levels are being checked before and after treatment. Subjects are requested to self-report their number of episodes or days of heroin use and 0-10-point visual analogue scale scores for heroin craving/refusal to use heroin during the previous week before and after treatment. Quality of life will be reported using the Short Form-12v2 before and after 4 weeks of treatment. Pulse diagnosis will be recorded and heart rate variability calculated before and after treatment. The baseline patient characteristics will be compared between the experimental and control groups using the independent t-test and chi-square test. Data are compared between the two groups using repeated-measures analysis of variance, generalized estimating equations, and the paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of OUD is confirmed using the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition. Subjects aged 20-70 years with OUD who have received methadone maintenance treatment for at least 1 month and provided informed consent are being recruited. Psychiatrists assess each prospective participant's eligibility to be enrolled in the study.

Exclusion Criteria:

* Subjects with a critical illness
* those who have taken Chinese herbs or received acupuncture treatment during the previous 30 days
* those who are unsuitable for recruitment in the opinion of the attending physician
* those who are unwilling to provide informed consent are excluded.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2024-02-14 (Estimated); Study Completion 2024-02-14 (Estimated)

PRIMARY OUTCOMES:
urinary morphine levels | 4 weeks
  morphine levels in urine
times or days of heroin use during the previous week | 4 weeks
  self-reported times or days of heroin use during the previous week

SECONDARY OUTCOMES:
self-reported visual analogue scale (VAS) scores for heroin craving/refusal to use heroin (0-10 points) in the previous week | 4 weeks
  A VAS score of 0 for heroin craving indicates no heroin craving and a score of 10 indicates the strongest possible heroin craving. A VAS score of 0 for refusal to use heroin indicates no refusal and a score of 10 indicates total refusal.
self-reported quality of life using the Short Form-12v2® | 4 weeks
  The PRO CoRE will be used to score the SF-12v2 Health Survey.
pulse diagnosis and heart rate variability | 4 weeks
  pulse diagnosis and heart rate variability will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Long Hu, MD, MS, Principal Investigator — Chief, Division of Acupuncture, Kaohsiung Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan